CLINICAL TRIAL: NCT00726245
Title: PRP as a Treatment for Acute Muscle Tears - Randomized-double-blind-placebo Control Trail.
Brief Title: Plasma Rich in Growth Factors (PRGF) Treatment for Muscle Tear
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Omer Mei-Dan, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3000
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Muscle Tear

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): PRGF
  Interventions: Biological: PRGF
- 2 (Placebo Comparator): physiological saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PRGF — 3-6mg IM (to area of muscle tear)
  Arms: 1
Biological: Placebo — 3cc IM of physiological saline
  Arms: 2

SUMMARY:
the improvement of symptoms and disease progress by the treatment of OA of the knee with PRGF

ELIGIBILITY:
Inclusion Criteria:

* US diagnosed muscle tear
* age 15-40 years old

Exclusion Criteria:

* pregnancy
* mental or physical disabilities

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
improvement of symptoms / disease progress | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medicak Center, Kfar Saba, Israel